CLINICAL TRIAL: NCT02360332
Title: A Collaborative Public/Private Employment Training and Placement Model for Transition Age Youth With Autism Spectrum Disorder (ASD)
Brief Title: A Collaborative Public/Private Employment Training and Placement Model ASD Transition Age Youth With Autism Spectrum Disorder (ASD)
Acronym: ProjSEARCH1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Henrico County Public Schools (Unknown); Virginia Department of Aging and Rehabilitative Services (Unknown); Chesterfield County Public Schools (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIDDRDRRP09-13
Record Dates: First submitted 2015-01-15; First posted 2015-02-10 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism; transition to adulthood; employment; High School Seniors
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PS-ASD (Experimental): Treatment Condition, participants assigned to this condition will receive the treatment, one school year (9 months) of Project SEARCH plus ASD Supports
  Interventions: Behavioral: Project SEARCH plus ASD Supports
- High School As Usual (No Intervention): Control Condition, Participants assigned to this condition will have no interaction or intervention with the research team with the exception of data collection at the specified time points.

INTERVENTIONS:
Behavioral: Project SEARCH plus ASD Supports — Project SEARCH program (Rutkowski, Daston, Kuiken, and Riehle, 2006) is a work based learning model for high school transition that was developed at Cincinnati Children's Hospital Medical Center. The model provides complete immersion in the workplace. Students spend their entire school day at the workplace for a full school year. Consistent with principles of work based learning, Project SEARCH facilitates the development of a broad range of high-quality jobs within the employer organization and provides over 700 of supervised work experience. The model also relies on the intensive application of supported employments strategies (task analysis and customization, systematic instruction, ongoing support, etc.) to allow the participation of individuals with extensive support needs.
  Other Names: PS-ASD
  Arms: PS-ASD

SUMMARY:
The aim of the research project is to conduct evidence-based research on a nationally known vocational rehabilitation (VR) service model (Project Search) for individuals with Autism Spectrum Disorders (ASD). This information may be useful to high schools and vocational rehabilitation agencies that endeavor to use evidence based practices to serve individuals with ASD.

DETAILED DESCRIPTION:
Autism is recognized to be a "complex disorder" as well as "a spectrum of disorders" that includes Asperger's syndrome and pervasive developmental disorder- not otherwise specified. Diagnostic criteria for autism focus on impairments affecting socialization, verbal and nonverbal communication, and restricted and repetitive patterns of behavior. The number of high school students diagnosed with autism, for example, has been increasing over time with almost 194,000 students ages 6 through 21 nationwide identified as having autism and receive special education services under the Individuals with Disabilities Education Act (IDEA). These young people create a significant need for vocational rehabilitation intervention in the decade ahead. Currently many persons with ASD continue to be. Howlin, et al. (2004) described the outcomes for 68 young adults with ASD (mean age 29), and found that a third worked and almost half were unemployed. RSA notes that in 2005 fewer than 2000 individuals with ASD received VR services. In Virginia the figure is only 255 total clients enrolled from between 2000 and 2007.

In this project the investigators will conduct a randomized clinical trial which examines the impact of intensive community-based work experiences on the employment outcomes of youth with ASD. This study will test the efficacy of a nationally recognized model of an employer based employment training and placement program (Project SEARCH) for youth with ASD. Four dependent measures will be investigated: (1) employment status upon completion of the program, at 90 days post completion and 12 months post completion (primary), (2) wage upon completion, at 90 days post completion, and 12 months post completion (secondary), (3) number of hours worked per week (secondary) upon completion, at 90 days post completion and 12 months post completion. Three specific hypotheses are proposed, and (4) intensity of supports needed at work at completion, at 90 days post completion and 12 months post completion.

Hypothesis I: Individuals who participate in an employer based employment training and placement program will demonstrate a higher rate of employment than those in the control condition.

Hypothesis II: Individuals who participate in an employer based employment training and placement program will earn higher wages on average at project completion compared to those in the control condition.

Hypothesis III: Individuals who participate in an employer based employment training and placement program will work more hours per week on average than those in the control condition.

Hypothesis IV: Individuals who participate in an employer based employment training and placement program will require less intensive work support than those in the control condition.

ELIGIBILITY:
Inclusion Criteria:

1. Being a student in the local public school where the research was being conducted,
2. Having an ASD medical diagnosis and/or educational eligibility,
3. Displaying independent self-care,
4. Being able to provide consent or assent,
5. Having funding for supported employment through VR, and
6. Having continued eligibility for public school educational services in the coming school year.

Exclusion Criteria:

1. Life threatening or dangerously severe aggressive or destructive behavior
2. History of fire setting
3. History of substance abuse

Ages: 18 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2009-10; Primary Completion 2013-09 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Change in Employment Status across 3 points in time (Employed or not employed) | 9 months, 12 months, 21 months
  Are subjects currently employed?

SECONDARY OUTCOMES:
Change in Hours worked weekly across 3 points in time | 9 months, 12 months, 21 months
  How many hours do subjects work weekly
Change in Hourly wage earned across 3 points in time | 9 months, 12 months, 21 months
  How much money do subjects earn hourly
Change in Intensity of work support required across 3 points in time | 9 months, 12 months, 21 months
  What type and how much do support do subjects require at work?

CONTACTS AND LOCATIONS:
Overall Officials: Paul Wehman, PhD, Principal Investigator — Virginia Commonwealth University

REFERENCES:
- [Background] Schall, C. M. (2010). Positive behavior support: Supporting adults with autism spectrum disorders in the workplace. Journal of Vocational Rehabilitation, 32, 109-115.
- [Background] Schall, C. M. & McDonough, J. T. (2010). Autism Spectrum Disorders in Adolescence and Early Adulthood: Characteristics and Issues. Journal of Vocational Rehabilitation, 32, 81-88.
- [Background] Schall C, Wehman P, McDonough JL. Transition from school to work for students with autism spectrum disorders: understanding the process and achieving better outcomes. Pediatr Clin North Am. 2012 Feb;59(1):189-202, xii. doi: 10.1016/j.pcl.2011.10.009. PMID 22284802
- [Background] Wehman, P., Schall, C., McDonough, J., Molinelli, A., Riehle, E., Ham, W., & Thiss, W. (2014). Project SEARCH for youth with autism spectrum disorders: Increasing competitive employment on transition from high school. Journal of Positive Behavior Intervention, 15, 144-155.
- [Background] Wehman, P., Schall, C., Carr, S., Targett, P., West, M., & Cifu, G., (2014). Transition from school to adulthood for youth with ASD: What we know and what we need to know. Journal of Disability Policy Studies, 25, 30-40; DOI: 10.1177/1044207313518071.
- [Background] Wehman PH, Schall CM, McDonough J, Kregel J, Brooke V, Molinelli A, Ham W, Graham CW, Erin Riehle J, Collins HT, Thiss W. Competitive employment for youth with autism spectrum disorders: early results from a randomized clinical trial. J Autism Dev Disord. 2014 Mar;44(3):487-500. doi: 10.1007/s10803-013-1892-x. PMID 23893098
- [Background] Ham, W., McDonough, J., Molinelli, A., Schall, C., & Wehman, P. (2014). Employment Supports for Young Adults with ASD: Two Case Studies. Journal of Vocational Rehabilitation. DOI: 10.3233/JVR-140677.
- [Derived] Wehman P, Schall CM, McDonough J, Graham C, Brooke V, Riehle JE, Brooke A, Ham W, Lau S, Allen J, Avellone L. Effects of an employer-based intervention on employment outcomes for youth with significant support needs due to autism. Autism. 2017 Apr;21(3):276-290. doi: 10.1177/1362361316635826. Epub 2016 Jul 9. PMID 27154907